CLINICAL TRIAL: NCT07257380
Title: Feasibility of Circulating Tumor DNA Based Minimal Residual Disease-Guided Adjuvant Therapy in Locally Advanced Gastric Cancer With Neoadjuvant Treatment: An Adaptive Trial (MRD-ATLAS)
Acronym: MRD-ATLAS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xuefei.Wang, Chief of Department of Gastrointestinal Surgery, Shanghai Zhongshan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-604R
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Gastric / Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric / Gastroesophageal Junction Adenocarcinoma; Circulating Tumor DNA; Minimal Residual Disease; Perioperative treatment
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Participants in this group will receive four cycles of neoadjuvant therapy followed by radical gastrectomy. Postoperatively, patients will be stratified based on their ctDNA MRD status at the post-surgical timepoint:
  1. ctDNA MRD-Negative Subgroup (estimated n=30): Patients will not receive adjuvant therapy (observation only).
  2. ctDNA MRD-Positive Subgroup (estimated n=30): Patients will receive adjuvant therapy.
  Interventions: Drug: Standard neoadjuvant therapy; Procedure: Radical gastrectomy; Drug: ctDNA-MRD-guided adjuvant therapy
- Control Arm (Active Comparator): This group serves as a standard-of-care comparison. Participants will receive four cycles of neoadjuvant therapy followed by radical gastrectomy. The decision to administer postoperative adjuvant therapy will be made by experienced clinicians based on standard treatment guidelines and the patient's individual condition.
  This group will include participants who meet any of the following criteria:
  1. Patients who decline ctDNA-guided postoperative adjuvant therapy strategies.
  2. Patients for whom insufficient tumor tissue was collected during screening to complete Whole Exome Sequencing (WES).
  3. Patients who are unwilling or unable to provide sufficient peripheral blood samples for ctDNA MRD testing.
  4. Any other conditions deemed unsuitable for inclusion in the Experimental Arm by the investigator.
  Interventions: Drug: Standard neoadjuvant therapy; Procedure: Radical gastrectomy; Drug: Standard adjuvant therapy

INTERVENTIONS:
Drug: Standard neoadjuvant therapy — Participants will receive 4 cycles of neoadjuvant therapy based on CSCO/NCCN guidelines. The specific regimen is determined by molecular characteristics and clinical practice:
  1. Chemotherapy: Options include SOX, DOS, FLOT, XELOX (CapeOx), or FOLFOX.
  2. HER2-Positive: Trastuzumab combined with chemotherapy, with or without immunotherapy.
  3. Immunotherapy: PD-(L)1 inhibitors may be administered as monotherapy or in combination with chemotherapy.
  Dosages and administration follow standard pharmaceutical labeling and institutional protocols.
Procedure: Radical gastrectomy — Radical gastrectomy with standard D2 lymphadenectomy will be performed.
Drug: Standard adjuvant therapy — Postoperative adjuvant therapy for the control group is determined by an experienced clinician based on standard clinical guidelines (e.g., CSCO, NCCN) and the patient's clinical status.
  The decision to administer adjuvant therapy, along with the specific regimen, is made at the discretion of experienced clinicians. If indicated, therapy typically begins 4-6 weeks post-surgery and consists of 4 cycles. The regimen generally mirrors the neoadjuvant therapy received and may include:
  1. Chemotherapy: Options include SOX, DOS, FLOT, XELOX (CapeOx), or FOLFOX.
  2. HER2-Positive: Trastuzumab combined with chemotherapy, with or without immunotherapy.
  3. Immunotherapy: PD-(L)1 inhibitors may be administered as monotherapy or in combination with chemotherapy.
  Dosages and administration follow standard pharmaceutical labeling and institutional protocols.
  Patients deemed unsuitable for adjuvant therapy by experienced clinicians will undergo observation.
  Arms: Control Arm
Drug: ctDNA-MRD-guided adjuvant therapy — Participants in the Experimental Arm will initially receive 4 cycles of neoadjuvant therapy followed by D2 radical gastrectomy. Postoperative management is strictly guided by ctDNA MRD status assessed at 4 weeks post-surgery:
  1. ctDNA MRD-Negative Subgroup: Participants will not receive adjuvant therapy and will undergo active surveillance (observation).
  2. ctDNA MRD-Positive Subgroup: Participants will receive 4 cycles of adjuvant therapy, initiating 4-6 weeks after surgery. The regimen generally mirrors the neoadjuvant therapy and is selected based on clinical guidelines (e.g., CSCO/NCCN). Options include: Chemotherapy: SOX, XELOX (CapeOx), FLOT, DOS, or FOLFOX . Targeted/Immunotherapy: Agents such as Trastuzumab (for HER2+) or PD-(L)1 inhibitors may be included if clinically indicated.
  Arms: Experimental Arm

SUMMARY:
Standard treatment for locally advanced gastric cancer currently involves surgery combined with chemotherapy administered both before and after the operation. However, post-surgery (adjuvant) chemotherapy often causes severe side effects, and it is unclear if all patients truly benefit from it. Recent research, such as the SPACE-FLOT study, suggests that patients who respond well to pre-surgery treatment might not actually benefit from further aggressive treatment after surgery; in these cases, additional therapy may only increase the risk of side effects without improving survival.

To address this, researchers are investigating circulating tumor DNA (ctDNA) testing, which detects microscopic traces of cancer (Molecular Residual Disease, or MRD) in the blood. The utility of ctDNA is supported by extensive research:

In Colorectal Cancer: The GALAXY study demonstrated that ctDNA status accurately predicts patient survival and identifies who benefits from chemotherapy. Furthermore, the DYNAMIC study showed that using ctDNA to guide treatment decisions significantly reduced the use of unnecessary chemotherapy without compromising patient survival.

In Gastric Cancer: Studies such as MENCA-GC, CRITICS, and PLAGAST have confirmed that post-surgery ctDNA is a strong predictor of patient prognosis. Additionally, the MRD-GATE study provided preliminary evidence that ctDNA-guided strategies can reduce unnecessary chemotherapy in the adjuvant setting.

Building on this evidence, this study applies ctDNA testing to the standard perioperative treatment model for gastric cancer. The primary objective is to determine if a ctDNA-guided strategy can identify patients who can safely forgo post-surgery chemotherapy, thereby reducing treatment toxicity and unnecessary usage, without sacrificing long-term survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide a written informed consent form (ICF), and understand, agree to, and comply with the study requirements and assessment schedule.
2. Male or female aged 18 to 79 years.
3. Histologically confirmed gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction (GEJ), with clinical TNM staging (per the 8th edition of the AJCC/UICC Clinical TNM Staging for Gastric Cancer) as clinical Stage cIII to cIVa, and the primary gastric cancer lesion assessed to be amenable to curative resection.
4. ECOG PS ≤ 2, tolerable to surgical treatment, no surgical contraindications.
5. Females of childbearing potential must have a negative pregnancy test within 7 days prior to initiating neoadjuvant treatment. Males of reproductive potential and females of childbearing potential must agree to use adequate contraceptive measures during the study and for 24 months after the last dose of study medication.
6. Prior to neoadjuvant treatment, complete blood count (CBC) and biochemical tests must meet the following criteria: a) Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L; b) Platelet Count (PLT) ≥ 75 × 10⁹/L; c) Hemoglobin (Hb) ≥ 80 g/L; d) Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × Upper Limit of Normal (ULN); e) Serum Creatinine (Cr) ≤ 1.5 × ULN, or Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73m²; f) Serum Albumin (ALB) ≥ 30 g/L; g) For subjects not receiving anticoagulant therapy: International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN, and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN; for subjects receiving anticoagulant therapy: PT value must be within the expected therapeutic range for the anticoagulant used.
7. No antitumor treatment for the tumor involved in the current study has been administered prior to the initiation of neoadjuvant treatment.

Exclusion Criteria:

1. Subjects for whom investigators consider that there are obvious contraindications to (neo)adjuvant treatment or who cannot tolerate (neo)adjuvant treatment.
2. Females of childbearing potential who have not undergone surgical sterilization or do not use adequate contraceptive measures, pregnant or lactating females, and males who plan to impregnate their partners in the near term.
3. Any severe or uncontrolled systemic disease, including but not limited to uncontrolled hypertension, active bleeding, diabetes mellitus, and others.
4. Severe chronic or active infections that require systemic antibacterial, antifungal, or antiviral therapy, including but not limited to tuberculosis (TB), human immunodeficiency virus (HIV) infection, and others.
5. History of previous malignant tumors or other malignant tumors currently present, except for basal cell or squamous cell skin cancer, superficial bladder cancer, prostatic/cervical/breast carcinoma in situ, and other such tumors that have been completely resected with no recurrence for at least 5 years.
6. Other circumstances that investigators deem inappropriate for study participation.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | From completion of adjuvant therapy (or radical gastrectomy for patients not receiving adjuvant therapy) up to 2 years, assessed every 3 months.
  RFS is defined as the time from the date of radical gastrectomy to the date of the first documented disease recurrence or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | From completion of adjuvant therapy (or radical gastrectomy for patients not receiving adjuvant therapy) up to 2 years, assessed every 3 months.
  OS is defined as the time from the date of radical gastrectomy to the date of death from any cause.
ctDNA Clearance Rate | Within 7 days prior to the initiation of neoadjuvant therapy. Within 7 days prior to radical gastrectomy. 3 to 5 weeks post-surgery. 4 weeks after completion of adjuvant therapy, or 5 months post-surgery.
  Defined as the proportion of patients whose ctDNA status converts from positive to negative.
The time point of ctDNA conversion from negative to positive and the time difference from the time point of radiological diagnosis of tumor recurrence | Within 7 days prior to radical gastrectomy. 3 to 5 weeks post-surgery. 4 weeks after completion of adjuvant therapy, or 5 months post-surgery.
  After peripheral blood collection, ctDNA detection is performed using a tumor-informed strategy based on NGS (Next-Generation Sequencing) and WES (Whole-Exome Sequencing) technologies.
Pathological Complete Response (pCR) Rate | Within 1 week after radical gastrectomy
  Pathological examination performed on gastric cancer surgical specimens

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, MD, PhD, Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai, China.
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No